CLINICAL TRIAL: NCT04987736
Title: Assessment of Long-term Effects (Complications) of COVID-19 in the Southern Part of Bangladesh - a Retrospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sher-E-Bangla Medical College (Other)
Responsible Party: Principal Investigator, Harendra Nath Sarker, Professor, Sher-E-Bangla Medical College
Other Study IDs: SBMC|Barisal|2020|1994
Record Dates: First submitted 2021-08-01; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: To Assess Long-term Effects of COVID-19 in Patients Who Were Affected With COVID -19
Keywords: long-term effects; COVID-19; RT-PCR +vE
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 (RT-PCR +ve) patients
  Interventions: Diagnostic Test: RT-PCR

INTERVENTIONS:
Diagnostic Test: RT-PCR — COVID 19 diagonostic test

SUMMARY:
An outbreak of the novel coronavirus nCoV-19 (SARS-CoV-2), responsible for the coronavirus disease-19 (COVID-19), was first detected in Hubei province, Wuhan, China, on December 31, 2019. It has rapidly spread globally with approximately 157,343,044 confirmed cases and 3,278,510 deaths till 7th May, 2021 [1]. World Health Organization (WHO) declared COVID- 19 pandemic on 11th March 2020.

The world is facing the second wave of Coronavirus Disease 2019 (COVID-19) pandemic which is the most troublesome challenge to public health. The second wave is running and nobody knows where we are in the course of this disease. It becomes a significant challenge for the public health, science, and medical sectors [2].

According to the World Health Organization, about 80% of infections are mild or asymptomatic, 15% result in moderate to severe symptoms (requiring oxygen) and about 5% are critical infections, which require ventilation.

We are learning something new every day. Our understanding of the pandemic is growing and changing daily. The world is focusing on the short term - flattening the curve, treating the sick and discovering a vaccine. But there is more to this pandemic than the short term.

We know a lot about the transmission and clinical feature of COVID-19, but relatively little about what happens after someone recovers. Much is still unknown about how COVID-19 will affect people over time. There's still much to be learned from those who have recovered from COVID-19.

DETAILED DESCRIPTION:
B. INTRODUCTION:

An outbreak of the novel coronavirus nCoV-19 (SARS-CoV-2), responsible for the coronavirus disease-19 (COVID-19), was first detected in Hubei province, Wuhan, China, on December 31, 2019. It has rapidly spread globally with approximately 157,343,044 confirmed cases and 3,278,510 deaths till 7th May, 2021 [1]. World Health Organization (WHO) declared COVID- 19 pandemic on 11th March 2020.

The world is facing the second wave of Coronavirus Disease 2019 (COVID-19) pandemic which is the most troublesome challenge to public health. The second wave is running and nobody knows where we are in the course of this disease. It becomes a significant challenge for the public health, science, and medical sectors [2].

According to the World Health Organization, about 80% of infections are mild or asymptomatic, 15% result in moderate to severe symptoms (requiring oxygen) and about 5% are critical infections, which require ventilation.

We are learning something new every day. Our understanding of the pandemic is growing and changing daily. The world is focusing on the short term - flattening the curve, treating the sick and discovering a vaccine. But there is more to this pandemic than the short term.

We know a lot about the transmission and clinical feature of COVID-19, but relatively little about what happens after someone recovers. Much is still unknown about how COVID-19 will affect people over time. There's still much to be learned from those who have recovered from COVID-19.

We are still only one year and four months beyond the first emergence of COVID-19, so it's too early to tell what the extent of any long-term impacts will be.

Most people who have COVID-19 recover completely within a few weeks [3]. But some people - even those who had mild disease, continue to experience symptoms after their initial recovery. Older people and people with many serious medical conditions like diabetes, COPD, heart disease, kidney disease etc. are the most likely to experience these lingering COVID-19 symptoms. The most common symptoms that linger over weeks, even months are:

* Fatigue
* Cough (dry)
* Shortness of breath
* Headache
* Joint pain
* Muscle pain
* Confusion and even hallucinations. But, our body has surprising healing capacity; most of these symptoms will improve by six months. However, some people recovering from COVID-19 will likely suffer from long-term health problems.

Although COVID-19 is seen as a disease that primarily affects the lungs, it can damage many other organs as well. This organ damage may increase the risk of long-term health problems. Some of the most common long-term effects are:

Lungs: The pneumonia associated with COVID-19 can often cause long-standing damage to the tiny air sacs (alveoli) in the lungs [4]. The resulting scar tissue i.e. pulmonary fibrosis can lead to long-term breathing problems.

Heart: A recent study from the University of Frankford in Germany showed abnormal heart findings in more than 75% of people studied who had recently recovered from COVID-19. Imaging tests taken months after recovery from COVID-19 have shown lasting damage to the heart muscle, even in people who experienced only mild COVID-19 symptoms. This may increase the risk of heart failure or other heart complications in the future.

Brain: COVID-19 can cause strokes [5], seizures and Guillain-Barre syndrome, even in young people. COVID-19 may also increase the risk of developing Parkinson's disease and Alzheimer's disease.

Blood clots and blood vessel problems: COVID-19 can predispose to form clots. While large clots can cause heart attacks and strokes, much of the heart damage caused by COVID-19 is believed to stem from very small clots that block tiny blood vessels (capillaries) in the heart muscle. Other organs affected by blood clots include the lungs, legs, liver and kidneys.

Psychiatric issues: Most people recovering from COVID-19 experience anxiety, depression, or cognitive impairment. Some may develop more serious Post-Traumatic Stress Disorder (PTSD) due to the trauma of the illness and treatment [6].

Kidney: Patient may develop kidney complications which could lead to a need for long-term dialysis.

A lot of things may happen in long run in those who recovered from COVID-19. Our understanding of COVID-19's long term effects will depend greatly on ongoing studies over the next decades.

C. OBJECTIVES:

1. General Objectives:

   To assess long-term effects of COVID-19 in patients who were affected with COVID -19 (RT-PCR +ve) from 1st July to 30th December, 2020 recorded in PCR Lab of Sher-E-Bangla Medical College Hospital, Barishal i.e. six months or more before the initiation of study and recovered fully.
2. Specific Objective:

To detect the system-based complications and assess their incidence, and compare the results with other studies in home and abroad.

D. METHODOLOGY:

Study Design: An observational retrospective study. Study Population: COVID -19 (RT-PCR +ve) patients from 1st July to 30th December, 2020 recorded in PCR Lab of Sher-E-Bangla Medical College Hospital, Barishal.

Inclusion Criteria:

* COVID-19 (RT-PCR +ve) patients age 20 years and above.
* Those patients whose mobile numbers are recorded in the register.
* Those patients who/their attendants are available on mobile phone.

Exclusion Criteria:

* Persons below 20 years of age.
* Those patients whose mobile numbers are not recorded in the register.
* Those patients who/their attendants are not available on mobile phone.
* Those who died by this time from causes unrelated to COVID-19.

Sample Size (n):

To determine the sample size the following formula was followed n= n= the desired sample size z= Standard normal deviate usually set at 1.96 p= Proportion in the population; if not known, it is regarded as 0.5 (50.0%), here p is 0.27 q= 1-p d= Degree of accuracy which is considered as 0.05 According to this formula the targeted sample was 302. But attempt will be taken to take more sample population as far as possible.

Sampling Technique:

Simple random sampling.

Place of Study:

Sher-E-Bangla Medical College Barishal Bangladesh.

Time-frame & Duration:

6 months from 1st July to 30th December 2021.

Research Instrument:

1. Record register of PCR lab
2. Printed questionnaire
3. Mobile phone
4. Prescription of registered doctor if any
5. Investigations if any.

Case definition:

1. Long-term effects of COVID-19 are those complications which develop or persist after 6 (six) months of COVID-19.
2. System-based complications should follow the standard definition and are listed in the questionnaire.

Statistical Analysis:

Statistical analyses will be carried out by using the Statistical Package for Social Sciences version 23 for Windows (SPSS Inc., Chicago, Illinois, USA). The mean and Standard deviation values will be calculated for continuous variables. t- test and analysis of variance (ANOVA) will be employed for continuous data. P values <0.05 was considered as statistically significant.

E. PROCEDURE:

The proposed study will be conducted in Sher-E-Bangla Medical College, Barishal, Bangladesh. Those who were RT-PCR positive for corona in PCR Lab of Sher-E-Bangla Medical College, Barishal from 1st July to 30th December, 2020 and recovered fully, will be listed from register of PCR Lab and their contact numbers will be collected from there. They will be contacted via cell phone and information will be collected after initial exchange of wellbeing and verbal consent. The conversation will be conducted by a registered physician as per prescribed questionnaire. If any complication is reported, then that will be confirmed either by the diagnosis of a registered physician (if already seen) or the patient will be advised to come and confirmed by respective specialist according to complication and specific investigation (if available). Follow-up will be done for at least 6 months after 6 months from the date of RT-PCR +ve by 3 telphonic conversation. All information will be registered in data collection form and analysed thereafter.

F. QUALITY CONTROL:

The quality control of this study will be supervised under the guidance of Professor Khan AK Azad, Ex. Principal, Professor and Head of the Department of Medicine, Dhaka Medical College, Dhaka under the SOP (Standard Operative Procedure).

G. INSTITUTIOAL APPROVAL:

We have already taken the institutional clearance from chairman, ethical committee, Sher-E-Bangla Medical College, Barishal, Bangladesh.

H. BUDGET:

Total Budget: BDT 3,50,000 (Approximately).

Detailed of the Budget:

Particulars BDT Doctor's salary- 1x6 months x 20000 120,000/- Data entry computer personel (Research associate's monthly salary 10000/-X 6) 60,000/= Specialist visit (Approximate) 40,000/= Investigations (Approximate) 1,00000/- Statistical analysis 15,000/= Stationary cost 10,000/= Others 5,000/= Total in Amount 3,50,000/=

I. FUNDING:

Contribution from researchers

J. OUTCOME:

At the end of study, we will be able to assess long-term effects of COVID-19 in patients of southern part of Bangladesh and to know its incidence. It will be possible to compare this with other studies in Bangladesh and other countries.

K. CONFLICTS OF INTEREST:

The investigator will not have any salary for himself from the fund. The salary will be provided to doctor, research associates and statistician.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 (RT-PCR +ve) patients age 20 years and above
* Those patients whose mobile numbers are recorded in the register
* Those patients who/their attendants are available on mobile phone

Exclusion Criteria:

* Persons below 20 years of age
* Those patients whose mobile numbers are not recorded in the register
* Those patients who/their attendants are not available on mobile phone
* Those who died by this time from causes unrelated to COVID-19

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COVID -19 (RT-PCR +ve) patients from 1st July to 30th December, 2020 recorded in PCR Lab of Sher-E-Bangla Medical College Hospital, Barishal.
Sampling Method: Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of long-term effects (complications) of COVID-19 in the southern part of Bangladesh | 6 Months
  At the end of study, we will be able to assess long-term effects of COVID-19 in patients of southern part of Bangladesh and to know its incidence.

CONTACTS AND LOCATIONS:
Locations (1):
- HN Sarker, Barishal, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
Decide later.

REFERENCES:
- [Result] WHO, Coronavirus disease 2019 (COVID-19) situation report, 7 May 2021, WHO Bull, 2021
- [Result] de Wit E, van Doremalen N, Falzarano D, Munster VJ. SARS and MERS: recent insights into emerging coronaviruses. Nat Rev Microbiol. 2016 Aug;14(8):523-34. doi: 10.1038/nrmicro.2016.81. Epub 2016 Jun 27. PMID 27344959
- [Result] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- See also: Related Info — https://www.mayoclinic.org/about-this-site/welcome
- See also: Related Info — https://www.hackensackmeridianhealth.org/HealthU/2020/05/20/can-covid-19-cause-a-stroke/
- See also: Related Info — https://www.nimh.nih.gov/health/topics/post-traumatic-stress-disorder-ptsd/